CLINICAL TRIAL: NCT04068415
Title: Development of a Constipation Risk Assessment Scale for Hospitalized Patients.
Acronym: ERCoPH
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/44
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Constipation
Keywords: Hospitalized patients
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Constipation risk assessment scale — questionnaires

SUMMARY:
Develop a risk assessment scale for constipation of hospitalized patients to identify at an early stage high-risk individuals and to implement the appropriate means of prevention.

DETAILED DESCRIPTION:
Constipation remains a prominent problem in the hospital care setting given the accumulation of contributing factors. Indeed, one of the most common causes of constipation is the existence of irregular habits in stool schedules, including the fact of delaying the time to go to the toilet, which causes the subject for a prolonged period of time to inhibit symptoms. defecation reflexes.

These disorders are often increased by the lack of exercise and prolonged bed rest, which cause a lack of muscle of the abdominal strap, the abdominals not being able to play their role of compression.

Some drugs are also a major cause of the difficulty of intestinal elimination, including opiates, anticholinergics, anti-depressants, etc.

Finally, an unbalanced diet, a water deficiency are aggravating factors, as is anxiety. In the medical and para-medical literature, there is no complete and validated tool for assessing the risk of constipation at the admission of a hospital stay. This project is to develop a constipation risk assessment scale, which can be used autonomously by nurses, based on the risk factors identified in the literature, scales published in English, and 2007 recommendations from the French National Society of Gastroenterology, recommendations of the High Authority of Health and a consensus of experts. The use of such a tool would make it possible to identify at an early stage high-risk individuals and to implement the appropriate means of prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Swallowing, drinking and eating
* Hospitalized in one of the participating services
* Hospitalized for a period of at least 4 days
* Able to give informed consent and answer questions about his or her lifestyle

Exclusion Criteria:

* Patient with major constipation at baseline (no stool for at least 6 days)
* History of intestinal surgery during the 10 days preceding the study,
* Hospitalized in palliative care or bed identified palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in services where constipation is a major concern : orthopedic surgery (Bordeaux), plastic surgery (Bordeaux), medical cardiology (Bordeaux) and internal medicine (Limoges).
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2012-05-06 (Actual); Primary Completion 2014-04-16 (Actual); Study Completion 2014-04-16 (Actual)

PRIMARY OUTCOMES:
Constipation yes/no | On the 4th day of hospitalization
  Less than a saddle in the first 4 days and prescription of laxatives

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BERGER, Mrs, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No